CLINICAL TRIAL: NCT06849154
Title: The Effectiveness of the REAL™, a School-based, Virtual Reality-integrated Social Emotional Learning Intervention to Promote Mental Health for Early Malaysian Adolescents
Acronym: REAL™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UKM PPI/111/8/JEP-2023-111; TRGS/1/2020/UKM/01/4/4 (Other Grant/Funding Number: Ministry of Education Malaysia)
Record Dates: First submitted 2025-02-16; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Anxiety; Depression Disorders; Emotional Regulation
Keywords: Adolescent mental health; Emotion regulation; School-based intervention; Virtual reality
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design, where participants are randomly assigned to either the intervention group, receiving the REAL™ module, or the control group, following the standard school curriculum. The intervention group undergoes structured sessions incorporating social-emotional learning (SEL) strategies and virtual reality (VR) components, while the control group receives no additional intervention. Outcomes are measured at four time points (baseline, immediate post-test, 3-month follow-up, and 6-month follow-up) to assess the effectiveness of the intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study used a single-blind design where participants and the outcomes assessor were initially masked to group assignments. Participants were not informed of their assignment at the beginning of the study to reduce expectancy effects. However, due to the nature of the intervention, participants eventually became aware of their group allocation. The outcomes assessor remained blinded throughout data collection and analysis, with all data coded to maintain objectivity and minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard School Curriculum (Control Group) (No Intervention): Participants in this group will continue with their usual school activities and will not receive the REAL™ Module intervention.
- REAL™ SEL Intervention Group (Experimental): Participants in this group will receive the REAL™ Module, a school-based social-emotional learning (SEL) intervention with virtual reality (VR).
  Interventions: Behavioral: REAL™ SEL Intervention Group

INTERVENTIONS:
Behavioral: REAL™ SEL Intervention Group — A structured intervention using virtual reality (VR) components to improve emotional regulation in early adolescents
  Arms: REAL™ SEL Intervention Group

SUMMARY:
The REAL™ (Read Emotions and Learn to Regulate) module is a school-based social-emotional learning (SEL) intervention designed for early adolescents in Malaysia. This study evaluates the effectiveness of the REAL™ intervention in improving emotional regulation skills and reducing depression and anxiety symptoms among secondary school students.

A randomized controlled trial (RCT) was conducted from February to November 2023, involving 226 students aged 13-14 years from four secondary schools in Selangor, Malaysia. The intervention integrates virtual reality (VR) components to enhance engagement and ensure that SEL skills are relatable within the students' sociocultural context.

Participants were assessed at four time points (baseline, immediate post-test, three-month follow-up, and six-month follow-up) using validated psychological measures, including the Difficulties in Emotion Regulation Scale (DERS), Beck Depression Inventory (BDI), and Beck Anxiety Inventory (BAI). The results showed that students in the intervention group demonstrated significant improvements in emotional regulation and reductions in depression and anxiety scores compared to the control group, with sustained benefits over time.

This study highlights the feasibility of implementing SEL programs in Malaysian schools and supports the integration of culturally adapted, VR-enhanced interventions to promote adolescent mental health.

DETAILED DESCRIPTION:
The REAL™ (Read Emotions and Learn to Regulate) module was developed as a school-based social-emotional learning (SEL) intervention designed to help early adolescents in Malaysia enhance their emotional regulation skills and reduce symptoms associated with depression and anxiety. Adolescence is a critical stage of emotional development, yet many young individuals struggle with managing their emotions effectively, which can impact their mental well-being and academic performance. While SEL programs have been widely implemented in various countries, culturally adapted interventions tailored to the Malaysian socio-cultural context remain limited. To address this gap, the REAL™ intervention integrates virtual reality (VR) components to enhance engagement and provide students with realistic, immersive experiences to practice emotion regulation strategies.

This study aims to evaluate the effectiveness of the REAL™ intervention in improving emotional regulation skills among lower secondary school students in Malaysia. A randomized controlled trial (RCT) was conducted from February to November 2023, involving 226 students aged 13-14 years from four secondary schools in Selangor, Malaysia. These schools were selected through multistage cluster sampling, and participants were randomly assigned to either the intervention group, which received the REAL™ SEL module, or the control group, which continued with the standard school curriculum.

The intervention consists of multiple sessions focusing on different aspects of SEL, including understanding emotions, identifying emotional triggers, cognitive restructuring, and applying regulation strategies in daily life. To reinforce learning, the intervention incorporates VR simulations that allow students to practice these skills in a controlled, interactive environment. This approach is designed to make SEL strategies more engaging, relatable, and effective for Malaysian adolescents.

Data collection occurs at four time points: baseline (T0), immediate post-test (T1), three-month follow-up (T2), and six-month follow-up (T3). The primary outcome measures include the Difficulties in Emotion Regulation Scale (DERS) for emotional regulation, the Beck Depression Inventory (BDI) for depressive symptoms, and the Beck Anxiety Inventory (BAI) for anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Malaysian citizens who are Form 1 and Form 2 students (ages 13-14).
2. Students who provide assent and obtain parental consent to participate.
3. Students enrolled in daily government secondary schools in Malaysia.
4. Students who can attend all four intervention sessions consecutively.

Exclusion Criteria:

1. Students from boarding-based schools, religious-based schools, or private schools.
2. Students with physical impairments that may hinder participation.
3. Students with intellectual deficits that may affect comprehension of the intervention.
4. Students diagnosed with severe mental illness.
5. Students currently receiving professional psychological treatment.

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 226 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Emotional Regulation Score | Baseline (T0), Immediate Post-Test (T1), 3-Month Follow-Up (T2), 6-Month Follow-Up (T3)
  : Measured using the Difficulties in Emotion Regulation Scale (DERS). Higher scores indicate greater difficulties in emotional regulation. A reduction in scores post-intervention suggests improved emotional regulation.

SECONDARY OUTCOMES:
Depression and Anxiety Scores | Baseline (T0), Immediate Post-Test (T1), 3-Month Follow-Up (T2), 6-Month Follow-Up (T3)
  Measured using the Beck Depression Inventory (BDI) for depression and Beck Anxiety Inventory (BAI) for anxiety. Higher scores indicate greater depressive and anxiety symptoms. A reduction in scores post-intervention suggests improvement in mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Nik Ruzyanei Nik Jaafar Prof. Dr., Master of Medicine Psychiatry, Study Director — Department of Psychiatry, Faculty of Medicine, Universiti Kebangsaan Malaysia (UKM)
Locations (1):
- Faculty of Medicine, Universiti Kebangsaan Malaysia (UKM), Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical considerations and privacy regulations regarding research involving minors.